CLINICAL TRIAL: NCT04889248
Title: Inspiratory Muscle Training in Respiratory Capacity, Heart Rate Variability, Life Quality and Emotional State in Patients With Amyotrophic Lateral Sclerosis.
Brief Title: Inspiratory Muscle Training With Powerbreath Device in Patients With ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ALS_UFV_21
Record Dates: First submitted 2021-05-14; First posted 2021-05-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Maximum Inspiratory Pressure; Diaphragm
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Inspiratory muscle training with Powerbreath IMT device, for a duration of 8 weeks. Treatment as usual
  Interventions: Other: Inspiratory Muscle Training with Powerbreath IMT device.
- Control (No Intervention): Without inspiratory muscle training. Treatment as usual.

INTERVENTIONS:
Other: Inspiratory Muscle Training with Powerbreath IMT device. — Inspiratory muscle training with Powerbreath IMT device, for a duration of 8 weeks.
  Each day, each subject perform 15 repetitions in the morning and evening, from Monday to Friday, resting on weekends.
  The endurance of the device increases along the study, initiating with the 30% of their own maximum inspiratory pressure (PImax) during the first week and increasing a 10% every other week, till reach the goal of 60% PImax.
  Arms: Intervention

SUMMARY:
Abstract:

Context/background: people affected by Amyotrophic Lateral Sclerosis (ALS) see their own life totally disturbed after the diagnosis. This disease also courses, apart from the functional and depressing worsening, with internal damage manifested by a cardio respiratory deterioration. There are not many clinical studies publications about this disease given that is considered a weird illness with short prognosis.

Objectives: to examine the effects of the inspiratory muscle training (IMT) on respiratory muscle strength, heart rate variability (HRV), quality of life and mood in patients with ALS.

Methods: 20 volunteer patients, male and female, with ALS, bulbar or spinal will take part of the cuasi-experimental study and they will be divided into two groups: an experimental group (n = 10) and a control group (n = 10). The Maximum Inspiratory Pressure (PIM), the HRV, the quality of life and mood will be measured. The participants of experimental group will conduct 30 inspirations per day, 15 in the morning and 15 in the evening, 5 days per week, through 8 weeks. The resistance of the training in the experimental group will be increase acording to the PIM measured at the first visit. During the first week, the resistance will be at 30% of PImax, weeks 2 and 3 at 40%, weeks 4 and 5 at 50% and the last 3 weeks at 60%. After 8 weeks, all participants will fill up again all scales and post training measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with ALS

Exclusion Criteria:

* PImax more than 30mmH2O
* Score higher than 2 in GDS Reisberg scale
* Using already respiratory devices during the day (except night CPAPs support) more than 14h/day.
* Unstable medical disease for the last 3 years.
* Use of IMT contraindicated for medical reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
PImax | 8 weeks
  Maximum Inspiratory Pressure

SECONDARY OUTCOMES:
HRV | 8 weeks
  Heart Rate Variability
HR | 8 weeks
  Heart Rate
ALSAQ-40 | 8 weeks
  The Amyotrophic Lateral Sclerosis Assessment Questionnaire
ALSFRS-R | 8 weeks
  ALS Functional Rating Scale Revised
Beck scale | 8 weeks
  Depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Davinia Vicente Campos, PhD, Principal Investigator — Universidad Francisco de Vitoria
Locations (1):
- Universidad Francisco de Vitoria, Pozuelo de Alarcón, Madrid, Spain